CLINICAL TRIAL: NCT04792190
Title: Use of Dapagliflozin to Reduce Burden of Atrial Fibrillation in Patients Undergoing Catheter Ablation of Symptomatic Atrial Fibrillation (DAPA-AF) Prospective, Randomized, Multicenter, Placebo-Controlled Trial
Brief Title: Use of Dapagliflozin to Reduce Burden of Atrial Fibrillation in Patients Undergoing Catheter Ablation of Symptomatic Atrial Fibrillation
Acronym: DAPA-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Mehmet Aktas, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00005844
Record Dates: First submitted 2021-01-29; First posted 2021-03-10 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Management Arm (Dapagliflozin) (Active Comparator): A block randomization method will be use to randomize subjects to treatment with dapagliflozin 10 mg once daily. Subjects will take 1 blinded tablet of study drug (dapagliflozin) dosed once daily, per the randomization scheme, for 12 months. Each subject will be dispensed 35 blinded doses per month, during each month of participation in the trial. Quarterly pill counts will be performed to track compliance.
  Interventions: Drug: dapagliflozin
- Control Arm (Placebo) (Placebo Comparator): Subjects will take 1 blinded tablet of placebo drug dosed once daily, per the randomization scheme, for 12 months. Each subject will be dispensed 35 blinded doses per month, during each month of participation in the trial. Quarterly pill counts will be performed to track compliance.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dapagliflozin — Subjects will take 1 blinded tablet of study drug (dapagliflozin 10 mg) dosed once daily, for 12 months.
  Arms: Intervention Management Arm (Dapagliflozin)
Drug: Placebo — Subjects will take 1 blinded capsule of placebo drug dosed once daily
  Arms: Control Arm (Placebo)

SUMMARY:
This is a multicenter trial to evaluate the impact of treatment with dapagliflozin versus placebo following catheter ablation of atrial fibrillation (AF) on the burden of AF during 6-12 months of follow-up. This prospective, randomized, multicenter, placebo-controlled trial aims to enroll 25 subjects with AF (paroxysmal or persistent) who are scheduled to undergo catheter ablation of patients.

DETAILED DESCRIPTION:
This is a multicenter trial to evaluate the impact of treatment with dapagliflozin versus placebo following catheter ablation of AF on the burden of AF during 6-12 months of follow-up. This prospective, randomized, multicenter, placebo-controlled trial aims to enroll 25 subjects with AF (paroxysmal or persistent) who are scheduled to undergo catheter ablation of patients. All enrolled subjects will be required to have a cardiac implantable electronic device (CIED) capable of assessing the burden of AF. Following catheter ablation for AF and functional CIED subjects will be randomized to treatment with dapagliflozin 10 mg once daily versus placebo. The primary endpoint for the trial will be AF burden assessed at 6-12 months following catheter ablation of AF. The Investigational Drug Services at the University of Rochester will be in charge of dispensing all study related drugs to subject.

ELIGIBILITY:
Inclusion Criteria

* Eligible for treatment with dapagliflozin per current FDA-approved indications, including: 1) heart failure (NYHA class II-IV) with reduced left ventricular ejection fraction (<50%), or 2) type 2 diabetes mellitus and established cardiovascular (CV) disease or multiple CV risk factors, or 3) as an adjunct to diet and exercise to improve glycemic control in adults with type 2 diabetes mellitus, 4) adults with chronic kidney disease at risk of progression as defined by the National Kidney Foundation as estimated GFR <60 ml/minute/1.73 m2.
* Scheduled to undergo ablation of symptomatic paroxysmal or persistent AF prior to date of randomization per current guideline indications.
* A glycated hemoglobin level < 10.5% during the past 6 calendar months prior to consent only in patients with type 2 diabetes mellitus
* Age > 18 years
* Existing functional CIED or planned to undergo CIED implant as SOC before or within 24 hours following the AF ablation procedure and prior to randomization date.

Exclusion Criteria

* Type 1 diabetes mellitus
* History of diabetic keto-acidosis
* Child Pugh Class C liver disease
* Last measured estimated GFR < 25 ml/minute/1.73 m2
* Pregnancy, plan to become pregnant <1 year after consent or breast feeding
* Current therapy with an SGLT2 inhibitor
* Hypersensitivity to dapagliflozin
* On heart transplant list or likely to undergo heart transplant
* Unwilling or unable to cooperate with the protocol
* Participation in other clinical trials (observational registries are allowed with approval).
* Unwilling to sign the consent for participation
* Life expectancy <1 year after consent date for any medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Aktas, MD, Principal Investigator — Principal Investigator
Locations (3):
- United States (3):
  - Maine Medical Center, Portland, Maine
  - Henry Ford Hospital, Detroit, Michigan
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Jackson SL, Tong X, Yin X, George MG, Ritchey MD. Emergency Department, Hospital Inpatient, and Mortality Burden of Atrial Fibrillation in the United States, 2006 to 2014. Am J Cardiol. 2017 Dec 1;120(11):1966-1973. doi: 10.1016/j.amjcard.2017.08.017. Epub 2017 Aug 30. PMID 28964382
- [Background] Patel NJ, Deshmukh A, Pant S, Singh V, Patel N, Arora S, Shah N, Chothani A, Savani GT, Mehta K, Parikh V, Rathod A, Badheka AO, Lafferty J, Kowalski M, Mehta JL, Mitrani RD, Viles-Gonzalez JF, Paydak H. Contemporary trends of hospitalization for atrial fibrillation in the United States, 2000 through 2010: implications for healthcare planning. Circulation. 2014 Jun 10;129(23):2371-9. doi: 10.1161/CIRCULATIONAHA.114.008201. Epub 2014 May 19. PMID 24842943
- [Background] Kim MH, Johnston SS, Chu BC, Dalal MR, Schulman KL. Estimation of total incremental health care costs in patients with atrial fibrillation in the United States. Circ Cardiovasc Qual Outcomes. 2011 May;4(3):313-20. doi: 10.1161/CIRCOUTCOMES.110.958165. Epub 2011 May 3. PMID 21540439
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Zimetbaum P. Antiarrhythmic drug therapy for atrial fibrillation. Circulation. 2012 Jan 17;125(2):381-9. doi: 10.1161/CIRCULATIONAHA.111.019927. No abstract available. PMID 22249528
- [Background] Gupta A, Perera T, Ganesan A, Sullivan T, Lau DH, Roberts-Thomson KC, Brooks AG, Sanders P. Complications of catheter ablation of atrial fibrillation: a systematic review. Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1082-8. doi: 10.1161/CIRCEP.113.000768. Epub 2013 Nov 15. PMID 24243785
- [Background] Freeman JV, Tabada GH, Reynolds K, Sung SH, Liu TI, Gupta N, Go AS. Contemporary Procedural Complications, Hospitalizations, and Emergency Visits After Catheter Ablation for Atrial Fibrillation. Am J Cardiol. 2018 Mar 1;121(5):602-608. doi: 10.1016/j.amjcard.2017.11.034. Epub 2017 Dec 14. PMID 29331355
- [Background] Deshmukh A, Patel NJ, Pant S, Shah N, Chothani A, Mehta K, Grover P, Singh V, Vallurupalli S, Savani GT, Badheka A, Tuliani T, Dabhadkar K, Dibu G, Reddy YM, Sewani A, Kowalski M, Mitrani R, Paydak H, Viles-Gonzalez JF. In-hospital complications associated with catheter ablation of atrial fibrillation in the United States between 2000 and 2010: analysis of 93 801 procedures. Circulation. 2013 Nov 5;128(19):2104-12. doi: 10.1161/CIRCULATIONAHA.113.003862. Epub 2013 Sep 23. PMID 24061087
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Hosseini SM, Rozen G, Saleh A, Vaid J, Biton Y, Moazzami K, Heist EK, Mansour MC, Kaadan MI, Vangel M, Ruskin JN. Catheter Ablation for Cardiac Arrhythmias: Utilization and In-Hospital Complications, 2000 to 2013. JACC Clin Electrophysiol. 2017 Nov;3(11):1240-1248. doi: 10.1016/j.jacep.2017.05.005. Epub 2017 Aug 2. PMID 29759619
- [Background] Frustaci A, Chimenti C, Bellocci F, Morgante E, Russo MA, Maseri A. Histological substrate of atrial biopsies in patients with lone atrial fibrillation. Circulation. 1997 Aug 19;96(4):1180-4. doi: 10.1161/01.cir.96.4.1180. PMID 9286947
- [Background] De Jong AM, Maass AH, Oberdorf-Maass SU, Van Veldhuisen DJ, Van Gilst WH, Van Gelder IC. Mechanisms of atrial structural changes caused by stretch occurring before and during early atrial fibrillation. Cardiovasc Res. 2011 Mar 1;89(4):754-65. doi: 10.1093/cvr/cvq357. Epub 2010 Nov 11. PMID 21075756
- [Background] Samman Tahhan A, Sandesara PB, Hayek SS, Alkhoder A, Chivukula K, Hammadah M, Mohamed-Kelli H, O'Neal WT, Topel M, Ghasemzadeh N, Ko YA, Aida H, Gafeer M, Sperling L, Vaccarino V, Liang Y, Jones DP, Quyyumi AA. Association between oxidative stress and atrial fibrillation. Heart Rhythm. 2017 Dec;14(12):1849-1855. doi: 10.1016/j.hrthm.2017.07.028. Epub 2017 Jul 27. PMID 28757307
- [Background] Wijffels MC, Kirchhof CJ, Dorland R, Allessie MA. Atrial fibrillation begets atrial fibrillation. A study in awake chronically instrumented goats. Circulation. 1995 Oct 1;92(7):1954-68. doi: 10.1161/01.cir.92.7.1954. PMID 7671380
- [Background] Wright EM, Loo DD, Hirayama BA. Biology of human sodium glucose transporters. Physiol Rev. 2011 Apr;91(2):733-94. doi: 10.1152/physrev.00055.2009. PMID 21527736
- [Background] Nauck MA, Del Prato S, Meier JJ, Duran-Garcia S, Rohwedder K, Elze M, Parikh SJ. Dapagliflozin versus glipizide as add-on therapy in patients with type 2 diabetes who have inadequate glycemic control with metformin: a randomized, 52-week, double-blind, active-controlled noninferiority trial. Diabetes Care. 2011 Sep;34(9):2015-22. doi: 10.2337/dc11-0606. Epub 2011 Aug 4. PMID 21816980
- [Background] Wilding JP, Woo V, Soler NG, Pahor A, Sugg J, Rohwedder K, Parikh S; Dapagliflozin 006 Study Group. Long-term efficacy of dapagliflozin in patients with type 2 diabetes mellitus receiving high doses of insulin: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):405-15. doi: 10.7326/0003-4819-156-6-201203200-00003. PMID 22431673
- [Background] Rosenstock J, Jelaska A, Frappin G, Salsali A, Kim G, Woerle HJ, Broedl UC; EMPA-REG MDI Trial Investigators. Improved glucose control with weight loss, lower insulin doses, and no increased hypoglycemia with empagliflozin added to titrated multiple daily injections of insulin in obese inadequately controlled type 2 diabetes. Diabetes Care. 2014 Jul;37(7):1815-23. doi: 10.2337/dc13-3055. Epub 2014 Jun 14. PMID 24929430
- [Background] Cavender MA, Norhammar A, Birkeland KI, Jorgensen ME, Wilding JP, Khunti K, Fu AZ, Bodegard J, Blak BT, Wittbrodt E, Thuresson M, Fenici P, Hammar N, Kosiborod M; CVD-REAL Investigators and Study Group. SGLT-2 Inhibitors and Cardiovascular Risk: An Analysis of CVD-REAL. J Am Coll Cardiol. 2018 Jun 5;71(22):2497-2506. doi: 10.1016/j.jacc.2018.01.085. PMID 29852973
- [Background] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Background] Zelniker TA, Bonaca MP, Furtado RHM, Mosenzon O, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Budaj A, Kiss RG, Padilla F, Gause-Nilsson I, Langkilde AM, Raz I, Sabatine MS, Wiviott SD. Effect of Dapagliflozin on Atrial Fibrillation in Patients With Type 2 Diabetes Mellitus: Insights From the DECLARE-TIMI 58 Trial. Circulation. 2020 Apr 14;141(15):1227-1234. doi: 10.1161/CIRCULATIONAHA.119.044183. Epub 2020 Jan 27. PMID 31983236
- [Background] Verma S. Potential Mechanisms of Sodium-Glucose Co-Transporter 2 Inhibitor-Related Cardiovascular Benefits. Am J Cardiol. 2019 Dec 15;124 Suppl 1:S36-S44. doi: 10.1016/j.amjcard.2019.10.028. PMID 31741439
- [Background] Ansary TM, Nakano D, Nishiyama A. Diuretic Effects of Sodium Glucose Cotransporter 2 Inhibitors and Their Influence on the Renin-Angiotensin System. Int J Mol Sci. 2019 Feb 1;20(3):629. doi: 10.3390/ijms20030629. PMID 30717173
- [Background] Li H, Shin SE, Seo MS, An JR, Choi IW, Jung WK, Firth AL, Lee DS, Yim MJ, Choi G, Lee JM, Na SH, Park WS. The anti-diabetic drug dapagliflozin induces vasodilation via activation of PKG and Kv channels. Life Sci. 2018 Mar 15;197:46-55. doi: 10.1016/j.lfs.2018.01.032. Epub 2018 Feb 1. PMID 29409796
- [Background] Lee TM, Chang NC, Lin SZ. Dapagliflozin, a selective SGLT2 Inhibitor, attenuated cardiac fibrosis by regulating the macrophage polarization via STAT3 signaling in infarcted rat hearts. Free Radic Biol Med. 2017 Mar;104:298-310. doi: 10.1016/j.freeradbiomed.2017.01.035. Epub 2017 Jan 26. PMID 28132924
- [Background] Bonnet F, Scheen AJ. Effects of SGLT2 inhibitors on systemic and tissue low-grade inflammation: The potential contribution to diabetes complications and cardiovascular disease. Diabetes Metab. 2018 Dec;44(6):457-464. doi: 10.1016/j.diabet.2018.09.005. Epub 2018 Sep 26. PMID 30266577
- [Background] Li C, Zhang J, Xue M, Li X, Han F, Liu X, Xu L, Lu Y, Cheng Y, Li T, Yu X, Sun B, Chen L. SGLT2 inhibition with empagliflozin attenuates myocardial oxidative stress and fibrosis in diabetic mice heart. Cardiovasc Diabetol. 2019 Feb 2;18(1):15. doi: 10.1186/s12933-019-0816-2. PMID 30710997
- [Background] Sato T, Aizawa Y, Yuasa S, Kishi S, Fuse K, Fujita S, Ikeda Y, Kitazawa H, Takahashi M, Sato M, Okabe M. The effect of dapagliflozin treatment on epicardial adipose tissue volume. Cardiovasc Diabetol. 2018 Jan 4;17(1):6. doi: 10.1186/s12933-017-0658-8. PMID 29301516
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Chen LY, Chung MK, Allen LA, Ezekowitz M, Furie KL, McCabe P, Noseworthy PA, Perez MV, Turakhia MP; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Stroke Council. Atrial Fibrillation Burden: Moving Beyond Atrial Fibrillation as a Binary Entity: A Scientific Statement From the American Heart Association. Circulation. 2018 May 15;137(20):e623-e644. doi: 10.1161/CIR.0000000000000568. Epub 2018 Apr 16. PMID 29661944
- [Background] Chiang CE, Naditch-Brule L, Murin J, Goethals M, Inoue H, O'Neill J, Silva-Cardoso J, Zharinov O, Gamra H, Alam S, Ponikowski P, Lewalter T, Rosenqvist M, Steg PG. Distribution and risk profile of paroxysmal, persistent, and permanent atrial fibrillation in routine clinical practice: insight from the real-life global survey evaluating patients with atrial fibrillation international registry. Circ Arrhythm Electrophysiol. 2012 Aug 1;5(4):632-9. doi: 10.1161/CIRCEP.112.970749. Epub 2012 Jul 11. PMID 22787011
- [Background] Pandey A, Kim S, Moore C, Thomas L, Gersh B, Allen LA, Kowey PR, Mahaffey KW, Hylek E, Peterson ED, Piccini JP, Fonarow GC; ORBIT-AF Investigators and Patients. Predictors and Prognostic Implications of Incident Heart Failure in Patients With Prevalent Atrial Fibrillation. JACC Heart Fail. 2017 Jan;5(1):44-52. doi: 10.1016/j.jchf.2016.09.016. PMID 28034376
- [Background] Thihalolipavan S, Morin DP. Atrial fibrillation and heart failure: update 2015. Prog Cardiovasc Dis. 2015 Sep-Oct;58(2):126-35. doi: 10.1016/j.pcad.2015.07.004. Epub 2015 Jul 17. PMID 26192885
- [Background] Hess PL, Healey JS, Granger CB, Connolly SJ, Ziegler PD, Alexander JH, Kowey PR, Ruff CT, Flaker G, Halperin JL, Hart RG, Lopes RD. The Role of Cardiovascular Implantable Electronic Devices in the Detection and Treatment of Subclinical Atrial Fibrillation: A Review. JAMA Cardiol. 2017 Mar 1;2(3):324-331. doi: 10.1001/jamacardio.2016.5167. PMID 28097334
- [Background] Passman RS, Weinberg KM, Freher M, Denes P, Schaechter A, Goldberger JJ, Kadish AH. Accuracy of mode switch algorithms for detection of atrial tachyarrhythmias. J Cardiovasc Electrophysiol. 2004 Jul;15(7):773-7. doi: 10.1046/j.1540-8167.2004.03537.x. PMID 15250860
- [Background] Solari D, Bertero E, Miceli R, Brunelli C, Ameri P, Canepa M. Methods, accuracy and clinical implications of atrial fibrillation detection by cardiac implantable electronic devices. Int J Cardiol. 2017 Jun 1;236:262-269. doi: 10.1016/j.ijcard.2016.12.189. Epub 2017 Jan 14. PMID 28143653
- [Background] Blomstrom-Lundqvist C, Gizurarson S, Schwieler J, Jensen SM, Bergfeldt L, Kenneback G, Rubulis A, Malmborg H, Raatikainen P, Lonnerholm S, Hoglund N, Mortsell D. Effect of Catheter Ablation vs Antiarrhythmic Medication on Quality of Life in Patients With Atrial Fibrillation: The CAPTAF Randomized Clinical Trial. JAMA. 2019 Mar 19;321(11):1059-1068. doi: 10.1001/jama.2019.0335. PMID 30874754
- [Background] Wechselberger S, Kronborg M, Huo Y, Piorkowski J, Neudeck S, Passler E, El-Armouche A, Richter U, Mayer J, Ulbrich S, Pu L, Kirstein B, Gaspar T, Piorkowski C. Continuous monitoring after atrial fibrillation ablation: the LINQ AF study. Europace. 2018 Nov 1;20(FI_3):f312-f320. doi: 10.1093/europace/euy038. PMID 29688326

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Management Arm (Dapagliflozin) | Control Arm (Placebo)
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Management Arm (Dapagliflozin) | Control Arm (Placebo) | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (12) | 67 (10) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Time Spent in Atrial Fibrillation
Description: For the primary endpoint of AF burden, defined as percentage of time spent in AF (i.e. amount of time spent in AF divided by the total amount of time a patient was monitored), the student's t-test will be used to statistically compare the placebo group vs. the active treatment group. This approach is subject to an examination of the distribution of the percent time in AF. AF data will be collected using a cardiac implantable electronic device (CIED).
  AF burden assessed at 6-12 months following catheter ablation of AF, defined as percentage of time spent in AF (i.e. amount of time spent in AF divided by the total amount of time a subject was monitored).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Intervention Management Arm (Dapagliflozin) | Control Arm (Placebo)
Number analyzed (Participants) | 12 | 13
percentage of time | 2.74 (6.31) | 5.85 (12.85)

2. Secondary Outcome: Rate of Health Care Utilization
Description: Rate of health care utilization (recurrent hospitalizations, unplanned office visits, need for emergency room visits)
Time Frame: 6-12 months
Measure: Number; unit: events
Groups:
- Intervention: Dapagliflozin treatment healthcare utilization at 12 months
- Control Arm: Control arm healthcare utilization at 12 months
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 12 | 13
events | 132 | 104

3. Secondary Outcome: Percentage of Participants Hospitalized for Heart Failure Post Catheter Ablation of AF
Time Frame: 6-12 months
Measure: Number; unit: percentage of participants
Groups:
- Intervention; Control Arm: Heart failure hospitalization at 12 months
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 12 | 13
percentage of participants | 0 | 0

4. Secondary Outcome: Mean Quality of Life Score Using the QualiTy-of-life (AFEQT) Questionnaire
Description: The AFEQT questionnaire is an AF-specific health-related quality of life questionnaire designed to be used in clinical research. The responses on the AFEQT are scored on a Likert scale, 1 = "Not at all…" to 7 = "Extremely". Scores range from 0 to 100. A score of 0 corresponds to complete disability and a score of 100 corresponds to no disability.
Time Frame: Final visit, approximately 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention; Control Arm: AFEQT Score at 12 months
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 3 | 3
score on a scale | 20.7 (8.8) | 15.4 (26.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Management Arm (Dapagliflozin) | Control Arm (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/13
Other Adverse Events (participants affected / at risk) | 6/12 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Management Arm (Dapagliflozin) (N=12) | Control Arm (Placebo) (N=13)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Management Arm (Dapagliflozin) (N=12) | Control Arm (Placebo) (N=13)
nausea (Gastrointestinal disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 0 | 1
hypoglycemia (Endocrine disorders) | 0 | 1
eye pain (Eye disorders) | 0 | 1
forgetfullness (Nervous system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study did not reach its enrollment goals and therefore was underpowered to detection a difference in

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT04792190/Prot_SAP_000.pdf